CLINICAL TRIAL: NCT04657783
Title: French National Cohort of People With Type 1 Diabètes: the SFDT1 Study
Brief Title: French National Cohort of People With Type 1 Diabetes
Acronym: SFDT1
Status: Recruiting | Type: Observational
Sponsor: Fondation Francophone pour la Recherche sur le Diabete (Other)
Collaborators: Société Francophone du Diabète (Other); Sanoia (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Eli Lilly and Company (Industry); Abbott Diabetes Care (Industry); Air Liquide Santé International (Industry); Novo Nordisk A/S (Industry); Sanofi (Industry); Insulet Corporation (Industry); DexCom, Inc. (Industry); Luxembourg Institute of Health (Other Government); Creapharm (Unknown); Medtronic (Industry); mylife Diabetes Care AG (Industry); LifeScan (Industry)
Responsible Party: Sponsor
Other Study IDs: SFDT1
Record Dates: First submitted 2020-09-30; First posted 2020-12-08 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 1; Cardiovascular Diseases; Hypoglycemia; Patient Participation
Keywords: type 1 diabetes; cardiovascular disease; glucose variability; hypoglycemia; quality of life; insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Cardiovascular Diseases; Hypoglycemia; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — We will look for an association between CV events and inflammation, oxidative stress markers in urine, saliva or plasma. At the end of the research, the samples can be used for subsequent analyses not foreseen in the original protocol that may be interesting in the context of the pathology according to the evolution of scientific knowledge, provided that the patient is not opposed, as indicated in the information / consent form.
  Hair will be used for research of drug exposure and toxin impregnation.
  After DNA samples extraction, genetic association analyses will be performed. DNA microarrays will be realised. Several types of analysis may be considered depending on the phenotype of interest and will be studied in the cohort . Lately, the strategy of "genome-wide polygenic score" showed its power to cluster groups of patients.
  Moreover, we can also consider rare genetic variants studies by exome or whole genome sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular (CV) diseases are the most frequent type 1 diabetes (T1D) complications. A recent epidemiological study showed that patients with T1D have a two-fold CV mortality risk, even in case of good glycemic control. In addition, it has been shown that patients with T1D with no traditional CV risk factors had about a 80% higher risk of cardiovascular event compared to non-diabetic individuals. This indicates that further modifiable risk factors in relation to CV mortality remain to be identified.

One of the candidates that could help to disentangle the factors associated with the increased CV mortality in T1D patients is glycemic variability which could contribute to diabetes complications. Indeed, severe hypoglycaemia, one of the most severe consequence of glycaemic variability, are associated with a higher mortality in patients with type 1 and type 2 diabetes.

In order to evaluate the relation between glycemic variability, insulin therapy modalities and CV risk as well as some other questions related to health determinants of T1D, we are building up a large observational, prospective, multi-centric cohort study of patients gathering 15,000 patients with T1D, age above 6 years old, to perform the following:

* Collecting clinical information
* Evaluating Glycemic variability (assessed by the coefficient of variation of glucose (CV) calculated from automatically downloaded continuous glucose monitoring data (CGM)
* Biobanking including plasma, DNA, urine, saliva and hair.
* Collecting patients' reported outcomes through auto-questionnaires (online questionnaires).
* Doing an active follow-up for a period of 10 years with an intermediate visit every 3 years.
* Passive follow-up: link to national Health data system (Système National de Données de Santé, SNDS) in order to exhaustively collect health events as death, CV events and hospitalizations (including severe hypoglycemia).

DETAILED DESCRIPTION:
1. STUDY DESIGN & TIMELINE

   1.1 Study design The SFDT1 is an real-life non-randomized multicentric prospective study with limited intervention (biobanking, patient questionnaires during visits, and a direct-to-patient electronic follow-up).

   1.2 Timeline Participants will be actively followed-up for 10 years, with both clinical visits every 3 years and a regular online follow-up in-between visits through the e-PRO.

   Inclusion period: 5 years Duration of participation for each patient: active follow-up for 10 years / Passive follow up: 30 yeards Total duration of the study: 35 years
2. SITES' PROFILE The minimum of 70 expected recruiting sites are divided into three categories including university hospital centres, general hospital centres, and private diabetologist offices linked to hospital centers.
3. SAMPLE SIZE The sample size calculation was performed based on our primary objective which is to identify new risk factors of MACE, beyond the traditional risk factors. The investigators based our calculation on a dichotomous outcome (MACE yes/no) with a design of an independent prospective cohort. The investigators expect the new risk factors to be associated with CV risk with a low to moderate magnitude, with relative risk between 1.10 and 1.50. Based on our most extreme assumption (RR=1.10) and with an overall probability of MACE events set to 0.25 (Circulation 135 , 1522-1531, 2017) for the unexposed group during the 30 year follow-up, a power set to 80%, an α risk of 5%, and the exposed group considered as the extreme quintile group of the exposure of interest (glycaemic variability for instance), the required minimal number of patients is 15080.

   The investigators finally decided to target the inclusion of 15000 patients with T1D.
4. STUDIED POPULATION 4.1 Inclusion Criteria Adults and children (age >= 6 years)

   Type 1 diabetes, defined as:

   Age at diagnosis of diabetes > 1 year and <= 35 years Insulin treatment initiated within the first 12 months following diabetes discovery Affiliation to the French social security scheme (RIPH-2 constraint) Ability to speak and read French Ability to give written informed consent 4.2 Non-inclusion Criteria Patient under guardianship or protection for vulnerable people
5. BIAS 5.1 Investigator selection bias All diabetology care centers will be informed by the SFD channels (newsletter, conference, etc.) in order to limit selection bias. Any center can propose to join the study and its application will be evaluated upon its clinical research quality standards, track records and this study's inclusion and logistic (biobank) capacity. The objective is to include patients treated in universities and non university public and private centers; as well as in private practices.

   In this study, the investigators will not include the minority of patients with T1D only followed by their general practitioner.

   5.2 Patient selection bias In the centers, all patients fulfilling the inclusion and non inclusion criteria will be proposed to participate to SFDT1.

   Some parts of the study (e-PRO, CGM device data, Biobank, genetic analyses) will be optional according to the choices of the patients, inducing bias. For example, the oldest patients or the ones with a lower digital literacy or without digital support will less frequently participate to e-PRO. Therefore, confounding factors, including age and socioeconomic factors, will be taken into consideration to interpret the results of the study.

   5.3 Information bias Direct-to-patient data forms are self-reported by patients. Therefore, their medical accuracy and quality could be lower than those provided only by physicians. On the other hand, this methodology based on PROs not only allows to access richer information (QoL, etc.), compared to methodologies usually reported in clinical trials, but also at a higher frequency.

   CGM devices are not used by all patients. Consequently, glucose level real-time monitoring will be missing for some patients. The investigators consider this choice as to be the closest as possible of real-life conditions. On the other hand, the investigators are technically ready to manage other data formats uploaded by investigators from new monitoring devices.
6. BENEFITS / RISKS Since the proposed study will be observational-like, no extra visit will be required and no additional data will be requested beyond the ones that are supposed to be collected in usual care.

6.1 Benefits The participating patients will be clearly informed that they will not benefit directly but will contribute to a research effort that could make an impact on T1D care in the following years.

6.2 Risks Patients will be followed in routine care. They will not run any interventional action beyond the biobank samples collection. However, this act is optional.

With the project being sponsored by a non profit organisation, requiring and managing a consequent amount of data, on a long term, it has been designed in a privacy-by-design perspective with strong data securities with the support of a specialised partner (SANOÏA), as to bring the highest privacy and personal data security to the participants.

Patients will be informed of their rights according to GDPR.

burden of the disease: Delivering monthly or even quarterly questions and/or validated forms to patients during a significant number of years could increase the perceived and psychological burden of the disease.

To manage this risk some actions are engaged: the patients' forms are actively sourced, tuned and tested during study conception with patients' associations involved; the patients actively confirm their participation to the e-PRO platform; the patients can switch off the invitation service that reminds them by email / SMS that he has forms to fill; the patients can revoke their participation to the study whenever they want to;

STUDY CONDUCT

1. SITES

   1.1 Sites Recruitment Prior to the start of the study, the investigators plan to contact all kinds of French diabetes point-of-care centers by email or mail to offer to join the study with the support of the French-speaking society of Diabetes.

   The investigators aim to include at least 70 sites. 1.2 Sites Activation This initiation will include a detailed review (20 minutes) of the protocol and study procedures.

   Each site will receive the investigator study file, which contains all regulatory documents, by post before the initiation visit.

   The study site initiations will be performed on site. Three centers initiation visits will be analysed during internal project meetings. Any adaptations in terms of content presented during the initiation visits will be evaluated.

   Following initiation, each center will be contacted by phone to follow-up on patient's recruitment.

   Each biobank capable center will receive SOPs and adequate tubes for biological sampling from patients for the biobank.

   The investigators of each site will be informed on the expected way of using CGM device web portals in the perspective of getting harmonised data.
2. PATIENTS INFORMATION

   All patients (or caregivers for children) matching the inclusion criteria and not matching exclusion criteria are invited to participate during the inclusion period.

   The investigator will give the patient a "patient information sheet" and obtain the patient's agreement through a written informed consent.
3. PATIENTS ENROLLMENT MODALITIES 3.1 Inclusion

   To guarantee for a smooth study execution and patient motivation, it is critical that the minimal set of information required to include a patient and activate its e-PRO portal be input in a timely manner by the investigator.

   Also, the investigators will separate the inclusion related data ("flash inclusion") and the baseline visit related data.

   The "flash inclusion" required data are: date of inclusion, age, gender, year of disease onset, name + e-mail adress + mobile number, Once this flash inclusion done, the platform: generates the Anonymous Patient_ID that will have to be reported in the "corresponding" table staying in the site in the format according to their practices; activates the e-PRO participation funnel, Some sites might prefer to use a "buffer" form in paper format. In this case they commit to fill the data online in less than 24 hours.

   3.2 Baseline visit Clinical examination The routine standardised set of physical measurements of the patient will be collected and recorded in a case report form from trained staff.

   CGM device web portal Investigators will check the appropriate data-sharing activation with their enrolled patients' CGM device web portal.

   Face to face questionnaires In addition to usual clinical examination, investigators or clinical research associates (CRAs) will use validated questionnaires or parts of them

   6.3.3 Biobank sample collection Once a participant is enrolled and has given his or her consent, a biological sample collection is set up.

   Trained staff will withdraw different biological samples (serum, plasma, hair, urine, saliva) from each participant. In children, the amount of blood collected will be adjusted to the patient's body weight.

   3.4 Participation to the e-PRO Investigators will collect email and mobile phone number of recruited patients. This information will be automatically and safely stored in a separate database and this will allow a robot to contact the patient to send "invitations" to fill their PRO forms online.

   A few minutes after inclusion, patients will receive an email with a unique URL. By clicking on this link, they will be asked to input a secure code (OTP) received on their mobile phone. By processing to this 2-channel authentication the investigators assure the patients' effective identity. At this step the patients define their own password to access to the e-PRO.

   If this procedure is not completed the patient will receive 3 reminders by email and SMS. In the absence of any validation within 2 weeks, the patient will be tagged as "not participant" to the e-PRO.
4. PATIENT FOLLOW-UP MODALITIES

   4.1 Visits in Site

   Routine visits will be proposed every three years (±0.5 years) during 10 years during the active follow-up of the study.

   Each visit is made of: Clinical examination and usual care visit data (i.e.: CGM data retrieved if patient has a CGM or laboratory results), Face to face questionnaires, Biological analysis (biobank) if specifically consented, with an additional specific consent for genetic analyses.

   4.2 Between visits, in a direct-to-patient way When the patient actively consents with the confirmation funnel described in 6.3.4 then he receives regular invitations to fill his online forms. An "invitation" is a digital message (SMS and email) to invite the patient to fill his or her online form.

   These data are around the following dimensions: sex life, life with the disease, treatment burden, QoL, nutrition, sleep quality.
5. END OF STUDY

   Data collection will end at the last follow-up visit of the last patient included, which should theoretically be after 35 years after the first included patient. The database will then be cleaned and frozen to initiate the final analysis phase.
6. BIOBANK Collection of blood, saliva, hair and urine will be attempted for each participant at baseline. Availability of these samples will be indicated in the e-CRF.

6.1 Blood Total amount of blood: 25 ml (below 2.5% of total blood volume) are collected in various preparations.

In children, the amount of blood collected will be adjusted to the patients' body weight.

It is not preferable to use heparin as an anticoagulant, as heparin may interfere with subsequent amplification of DNA by PCR.

6.2 Urine One 5 ml tube will be collected and stored at -80°C.

6.3 Saliva Saliva sample is stable at ambient temperature but will be stored at -80°C.

6.4 Hair Hair will be used for research of drug exposure and toxin impregnation.

6.5 Storage All collected samples will be stored following regulatory conservation conditions (-80°C).

6.6 Circuit

UHC and GHC will collect the full complement of biological samples and will store them in regulatory conditions before sending them to the central laboratory.

Regular shipments (every 6 months):

1. at Creapharm
2. sending a sample to the laboratory of Lille for DNA extraction (genetic analysis)

6.6.7 Genetic analyses For participants (and caregivers for paediatric patients) who consented to do genetic analyses, DNA extraction will be done from blood samples.

Justification of genetic analysis : DNA microarrays will be realised. Several types of analysis may be considered depending on the phenotype of interest and will be studied in the cohort. Lately, the strategy of "genome-wide polygenic score" showed its power to cluster groups of patients. Moreover, the investigators can also consider rare genetic variants studies by exome or whole genome sequencing.

ELIGIBILITY:
1. Inclusion Criteria

   * Adults and children (age >= 6 years)
   * Type 1 diabetes, defined as:
   * Age at diagnosis of diabetes > 1 year and <= 35 years
   * Insulin treatment initiated within the first 12 months following diabetes discovery
   * Affiliation to the French social security scheme (RIPH-2 constraint)
   * Ability to speak and read French
   * Ability to give written informed consent
2. Non-inclusion Criteria Patient under guardianship or protection for vulnerable people

Ages: 6 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals leaving with type 1 diabètes, 6 years old or older
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2025-06-10 (Estimated); Study Completion 2035-06-10 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 30 years
  The MACE will include non-fatal myocardial infarction (MI), non-fatal stroke, and CV-related death (defined as a death occurring within 30 days after a diagnosis for MI, stroke, unstable angina, heart failure, sudden cardiac arrest, cardiogenic shock, other cerebrovascular events, or other CV events recorded in a medical claim in any setting).

SECONDARY OUTCOMES:
Non-fatal myocardial infarction (MI) | 30 years
  Defined from ICD-9-CM (430.xx, 431.xx, 434.xx, 436.xx) and ICD-10 CM (I60.xx, I61.xx, I63.3-I63.9, I66.xx)
CV-related death | 30 years
  Death secondary to following conditions :
  Myocardial infarction ICD-9-CM : 410.xx ICD-10 CM : I21.xx, I22.xx Stroke ICD-9-CM: 430.xx, 431.xx, 434.xx, 436.xx ICD-10 CM : I60.xx, I61.xx, I63.3-I63.9, I66.xx Unstable angina ICD-9-CM: 411.1x ICD-10 CM : I20.0 Congestive heart failure ICD-9-CM : 428.0x ICD-10 CM : I50.9 Other CVD-related conditions Sudden cardiac arrest ICD-9-CM : 427.5 ICD-10 CM : I46.9 Heart failure ICD-9-CM: 428.xx ICD-10 CM : I50.xx Cardiogenic shock ICD-9-CM: 785.51 ICD-10 CM : R57.0 Other cerebrovascular events ICD-9-CM : 432.xx, 433.xx, 435.xx, 437.xx ICD-10 CM : I62.xx, I63.0-I63.2, I65.xx, I67.xx, I68.xx Other cardiovascular events ICD-9-CM : 411.xx-414.xx, 415.xx-417.xx, 420.xx-427.xx, 429.xx ICD-10 CM : I20.x, I23.xx-I25.xx, I26.xx-I28.xx, I30.xx-I49.x, I51.xx-I52.xx, I64.xx
diabetic retinopathy without macumar edema | 30 years
  Defined from ICD-10-CM : E10.319
diabetic retinopathy with macular edema | 30 years
  Defined from ICD-10-CM : E10.311
diabetic nephropathy | 30 years
  Defined from ICD-10-CM : E10.21
All cause mortality | 30 years
  Mortality

CONTACTS AND LOCATIONS:
Locations (1):
- FFRD, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aguayo GA, Martin VP, Canha D, Cosson E, Arnault G, Delenne B, Guerci B, Berot A, Barraud S, Riveline JP, Fagherazzi G. Psychosocial burden in type 1 diabetes: a cross-sectional network analysis in the SFDT1 study. BMJ Open. 2026 Jan 29;16(1):e105713. doi: 10.1136/bmjopen-2025-105713. PMID 41611462
- [Derived] Canha D, Choudhary P, Cosson E, Banu I, Barraud S, Valero R, Ronci N, Delenne B, Dufaitre L, Vidal-Trecan T, Schaepelynck P, Sanz C, Tatulashvili S, Aguayo GA, Fagherazzi G, Riveline JP. Time below range alone is insufficient to identify severe hypoglycaemia risk in type 1 diabetes-the critical role of hypoglycaemia awareness: results from the SFDT1 study. Diabetologia. 2025 Dec;68(12):2719-2731. doi: 10.1007/s00125-025-06536-x. Epub 2025 Sep 9. PMID 40924111
- [Derived] Canha D, Aguayo G, Cosson E, Vaduva P, Renard E, Alzaid F, Bonnet F, Hadjadj S, Potier L, Verges B, Lablanche S, Benhamou PY, Hanaire H, Reznik Y, Riveline JP, Fagherazzi G. Clinical phenotyping of people living with type 1 diabetes according to their levels of diabetes-related distress: results from the SFDT1 cohort. BMJ Open Diabetes Res Care. 2025 Feb 24;13(1):e004524. doi: 10.1136/bmjdrc-2024-004524. PMID 40000027
- Available data/document: Study Protocol — https://drive.google.com/drive/my-drive